CLINICAL TRIAL: NCT04768725
Title: A Randomized Controlled Trial Investigating the Effects of Combined Physical-cognitive Exercise and Dietary Intervention on Cognitive Performance and Changes in Blood Biomarkers of Postmenopausal Obese Women
Brief Title: Combined Physical-cognitive Exercise and Dietary Intervention for Postmenopausal Obese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Somporn Sungkarat, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AMS-PT CMU 2564
Record Dates: First submitted 2021-02-05; First posted 2021-02-24 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Obesity
Keywords: Dietary intervention; Cognitive function; Brain-derived neurotrophic factor; Exergaming; Obesity
MeSH Terms: conditions — Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary intervention (Active Comparator): Participants will consume a self-selected diet with 25-75% of estimated baseline energy requirements for 2 days/week (fast day) along with ad libitum for 5 days/week (feed day).
  Interventions: Behavioral: Dietary intervention
- Physical-cognitive intervention (Active Comparator): Participants will perform home-based physical-cognitive training for 60 minutes per session, 3 session a week.
  Interventions: Behavioral: Physical-cognitive intervention
- Physical-cognitive with dietary intervention (Experimental): Participants will receive both dietary intervention and physical-cognitive training same as those in the dietary and physical-cognitive intervention groups.
  Interventions: Behavioral: Dietary intervention combined with physical-cognitive exergaming
- Control (No Intervention): Participants in the control group will be encouraged to continue their activities and calorie intakes as they usually would.

INTERVENTIONS:
Behavioral: Dietary intervention combined with physical-cognitive exergaming — Intermittent Fasting (IF) [self-selected diet with 25-75% of estimated baseline energy requirements for 2 days/week (fast day) along with ad libitum for 5 days/week (feed day)] combined with physical-cognitive exercise [60-70% of heart rate maximum for aerobic and 60-70% of 1 repetition maximum, 8-12 repetitions/set, 3 sets of each exercise for resistance exercise; memory, attention, and executive function for cognition], 60 minutes per session, 3 sessions per week for 12 weeks (36 sessions)].
  Arms: Physical-cognitive with dietary intervention
Behavioral: Dietary intervention — Intermittent Fasting (IF) [self-selected diet with 25-75% of estimated baseline energy requirements for 2 days/week (fast day) along with ad libitum for 5 days/week (feed day)].
  Arms: Dietary intervention
Behavioral: Physical-cognitive intervention — Physical-cognitive exercise [60-70% of heart rate maximum for aerobic and 60-70% of 1 repetition maximum, 8-12 repetitions/set, 3 sets of each exercise for resistance exercise; memory, attention, and executive function for cognition], 60 minutes per session, 3 sessions per week for 12 weeks (36 sessions)].
  Arms: Physical-cognitive intervention

SUMMARY:
This study aims to examine the effects of dietary intervention combined with physical-cognitive exergaming on cognitive performance and circulating biomarkers of obese postmenopausal women. It is hypothesized that participants will demonstrate significant improvement in cognitive performance and circulating biomarkers after participating in this combined program compared to baseline and the dietary and control groups.

DETAILED DESCRIPTION:
An association between obesity and cognitive impairment has been consistently reported. The risk of having dementia in later life is about 74% higher for middle-aged obese individuals than those with normal BMI. Estrogen deprivation has also been found to impair cognition. Thus, obese postmenopausal women are likely to be at risk of having cognitive impairment. The common recommendation for obesity management is dietary and exercise intervention. Research evidence has demonstrated that either dietary intervention or moderate-vigorous intensity exercise enhance cognitive function in obese adults. This study aims to examine the effects of 12-week home-based dietary intervention combined with physical-cognitive exergaming on cognitive performance and circulating biomarkers of obese postmenopausal women through a randomised controlled trial. Participants will be randomly assigned to one of the four groups: 1) dietary intervention 2) combined physical-cognitive exergaming, 3) dietary intervention combined with physical-cognitive exergaming, and 4) control group. Outcome measures including cognitive performance (i.e. executive function, episodic memory, attention, language, and global cognition), circulating biomarkers (i.e. BDNF level, metabolic parameters, inflammation markers, and adiponectin levels) as well as physical performance will be determined at baseline and after 12-week intervention. Findings from this study may offer a feasible and effective intervention program to improve cognitive performance along with its responsible circulating biomarkers in obese postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* obese women (body mass index (BMI) ≥ 25 kg/m2 with waist-to-hip ratio (WHR) ≥ 0.80)
* post-menopausal (self-reported menstrual characteristics (last menstruation > 1 year) or confirmed by blood follicular stimulating hormone (FSH) level ( > 20 IU/L) and estradiol level ( ≤ 30 pg/ml))
* sedentary lifestyle (exercise < 1 hr./wk.)
* normal range of the Mental State Examination T10 (MSET10) score
* at least 6 years of education
* own a mobile phone that supports application platform
* able to comply with the study schedule and procedures

Exclusion Criteria:

* have medical conditions that would be unsafe to exercise or have been diagnosed with neurological conditions (e.g. Parkinson's disease, stroke, multiple sclerosis) that affect cognition and mobility
* have weight variation ( > 5 kilogram in 3 months)
* have other dietary restrictions (e.g. vegetarianism and veganism)
* have depressive symptoms defined as a score ≥ 11 on Hospital Anxiety Depression Scale (HADS)
* have an uncorrected visual or hearing impairment
* receive hormonal replacement therapy

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2022-12-05 (Actual)

PRIMARY OUTCOMES:
change from baseline time to complete Trail Making B-A at 12 weeks | 12 weeks
  Time to complete Trail Making B and A will be recorded in seconds. The difference between time to complete Trail B and A will be used to index the task switching ability, a subdomain of executive function. Smaller differences between B-A indicate better switching ability.
change from baseline Stroop Color and Word score at 12 weeks | 12 weeks
  In Stroop Color and Word test, the number of items correctly identified in 45 seconds in each condition (i.e. word, color, color-word) will be recorded. Then the predicted score will be calculated. Score will be obtained from the different between the color-word and predicted scores. Lower scores indicate greater difficulty in inhibiting interference.
change from baseline Logical Memory score at 12 weeks | 12 weeks
  In Logical Memory test, participants will be instructed to listen carefully to two stories and remember their contents. After a 30-delay, they will be asked to freely recall the passages (recall) and respond yes or no to the given questions (recognition). The possible scores are 0-75. Higher scores indicate better episodic memory.
change from baseline Brain-derived neurotrophic factor (BDNF) level at 12 weeks | 12 weeks
  Level of plasma BDNF will be determined before and after the intervention.

SECONDARY OUTCOMES:
change from baseline Montreal Cognitive Assessment (MoCA) score at 12 weeks | 12 weeks
  The Montreal Cognitive Assessment will be used to index global cognitive function. The possible scores are 0-30. Higher scores indicate better cognitive function.
change from baseline Verbal Fluency score at 12 weeks | 12 weeks
  Category fluency subtest (naming test) of Verbal Fluency will be used. Participants will be asked to produce as many words as possible in 60 seconds. Higher scores indicate better language ability.
change from baseline Digit Span score at 12 weeks | 12 weeks
  In Digit Span test, lists of numbers will be presented orally to participants. They are asked to repeat the numbers immediately in ascending (forward) or reverse (backward) numerical order. The possible scores are 0-28. Higher scores indicate better attention.
change from baseline plasma adiponectin levels at 12 weeks | 12 weeks
  Level of plasma adiponectin will be determined before and after intervention.
change from baseline plasma Interleukin 6 (IL-6) levels at 12 weeks | 12 weeks
  Level of plasma IL-6 will be determined before and after intervention.
change from baseline insulin resistance levels at 12 weeks | 12 weeks
  Level of insulin resistance will be assessed using the homeostasis model assessment (HOMA-IR) index [fasting glucose (mg/dL) X fasting insulin (µU/mL) / 405].
change from baseline Six-minute walk distance at 12 weeks | 12 weeks
  The distance (in meters) participants walked in 6 minutes will be determined. Longer distance indicates better cardiorespiratory fitness.
change from baseline 30 seconds Chair Stand Test at 12 weeks | 12 weeks
  The number of repetitions participants could perform sit-to-stand will be recorded. Higher number of repetitions indicates greater lower-body strength.

CONTACTS AND LOCATIONS:
Overall Officials: Somporn Sungkarat, PhD, Principal Investigator — Chiang Mai University
Locations (1):
- Department of Physical Therapy, Faculty of Associated Medical Sciences, Chiang Mai University, Chiang Mai, Thailand

REFERENCES:
- [Derived] Keawtep P, Sungkarat S, Boripuntakul S, Sa-Nguanmoo P, Wichayanrat W, Chattipakorn SC, Worakul P. Effects of combined dietary intervention and physical-cognitive exercise on cognitive function and cardiometabolic health of postmenopausal women with obesity: a randomized controlled trial. Int J Behav Nutr Phys Act. 2024 Mar 5;21(1):28. doi: 10.1186/s12966-024-01580-z. PMID 38443944